CLINICAL TRIAL: NCT00364221
Title: The Effect of Rosiglitazone on Adipocyte-derived Cytokines in Nondiabetics With the Metabolic Syndrome
Brief Title: Effect of Rosiglitazone in Nondiabetic Patients With the Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-0447
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Metabolic Syndrome; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
The metabolic syndrome is a collection of health risks that includes obesity, high blood pressure, high triglycerides, high blood sugar, low good cholesterol, and resistance to insulin. The purpose of this study is to find out if the medication, rosiglitazone, influences levels of fat cell proteins and alters insulin resistance in nondiabetic persons with the metabolic syndrome. This is an early step to see if a medication, such as rosiglitazone, will be beneficial in people who have the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Nondiabetic subjects with an NCEP/ATP III diagnosis of the metabolic syndrome

Exclusion Criteria:

* Statin Medications, liver disease, cardiovascular disease, heart failure, diabetes, chronic kidney disease,

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-11; Primary Completion 2006-07 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Aquilante, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center General Clinical Research Center, Denver, Colorado, United States